CLINICAL TRIAL: NCT07092644
Title: Preeclampsia e Malformazioni Cardiache Fetali: Uno Sguardo al Cuore Materno
Brief Title: Preeclampsia and Fetal Heart Malformations: Looking to Maternal Heart
Acronym: MAMAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Salvi Silvia, Medical Doctor Specialised in Obstetrics and Gyanecology, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7552; Ethic Committee Gemelli (Other: 7552)
Record Dates: First submitted 2025-06-30; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Congenital Heart Disease
Keywords: Preeclampsia; Congenital Heart Disease; Maternal Hemodynamic
MeSH Terms: conditions — Heart Defects, Congenital; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodynamic evaluation in pregnant women carring a fetus with a congenital heart desease (Other): Hemodynamic indices will be obtained using the USCOM® system. Women will undergo a hemodynamic investigation at the time of first diagnosis of congenital heart disease during pregnancy or at the first assessment in Fondazione Policlinico A. Gemelli during pregnancy and then every two weeks until delivery. An additional hemodynamics evaluation will be performed in the post-partum period (in the 72 hours immediately after delivery). All hemodynamic assessment will be performed under standardized conditions.
  Interventions: Device: UltraSonic Cardiac Output Monitor (USCOM®)

INTERVENTIONS:
Device: UltraSonic Cardiac Output Monitor (USCOM®) — Using USCOM, the haemodynamic evaluation will be performed at the time of diagnosis of congenital heart desease and then every two weeks until delivery. A further evaluation will be performed immediately after delivery (within 72 hours).

SUMMARY:
The goal of this study is to describe the maternal hemodynamic parameters detected by UltraSonic Cardiac Output Monitor (USCOM®) in women carrying a fetus with a congenital heart disease (CHD) and to possibly describe an association between those parameters and the presence of a fetal cardiac anomaly.

It will also learn about:

* the number of cases of preeclampsia in our population of women carrying fetuses with CHD
* the relationship between maternal hemodynamic profile and maternal and perinatal outcome
* the associations between maternal hemodynamic parameters and the specific heart defect subtype
* the relationship between maternal hemodynamic parameters and fetal cardiac parameters in our population.

The haemodynamic evaluation will be performed at the time of diagnosis of CHD and then every two weeks until delivery. A further evaluation will be performed immediately after delivery (within 72 hours).

DETAILED DESCRIPTION:
The following maternal hemodynamic indices will be evaluated: heart rate (HR) (beats per min; bpm), mean arterial pressure (mmHg), stroke volume (mL), cardiac output (CO) (L/min), systemic vascular resistance (dynes/s/cm5). Data on the demographic and pregnancy characteristics of participants, hemodynamic and ultrasound investigations, perinatal and delivery features will be also collected. In particular, the following variables will be included in the study: type of congenital heart defect, gestational age at diagnosis, fetal weight (EFW) and fetal weight centile at diagnosis of CHD and at the last scan before delivery, mean uterine arteries pulsatility index (UtA-PI), fetal umbilical artery (UA-PI) and middle cerebral artery pulsatility index (MCA-PI) at diagnosis and at the last scan before delivery, maternal age, height, pre-pregnancy weight and gestational weight gain, systolic and diastolic blood pressure values (maximum and minimum values), presence of proteinuria, biochemical maternal assessment (maximun and miminum values of creatinine and uric acid level, platelet count, liver enzyme level), incidence of hypertensive disorders of pregnancy, antihypertensive drug administration (type and dosage) including magnesium sulfate, antenatal steroid administration, mode of delivery and indications, gestational age at delivery, birthweight and birthweight centile, need of respiratory or cardiac support, neonatal intensive care unit admission and number of days, major neonatal complications, maternal morbidities (HELLP, eclampsia, intravascular disseminate coagulation, post-partum hemorrhage), and mortality. The following definitions of hypertensive disorders will be used, according to the International Society for the Study of Hypertension in Pregnancy (ISSHP) 2018 criteria (14): chronic hypertension (CH) will be defined as hypertension (≥140/90mmHg) that predates pregnancy or is present prior to 20 weeks' gestation; gestational hypertension was defined as de-novo hypertension (≥ 140/90 mmHg) after 20 weeks' gestation; and preeclampsia (PE) will be defined as de-novo hypertension (≥ 140/90 mmHg) after 20 weeks' gestation with coexisting proteinuria, other maternal organ dysfunction or fetal growth restriction; preeclampsia superimposed to chronic hypertension (PE-CH).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent accepted
* Maternal Age ≥ 18 years
* Singleton pregnancy with a viable fetus at >20 weeks of gestation, with a diagnosis of congenital heart disease detected on antenatal ultrasound assessment and postnatally confirmed

Exclusion Criteria:

* Multiple pregnancy
* Pregnancy complicated by aneuploidy, genetic syndrome, or major structural fetal abnormality
* Maternal congenital heart disease (GUCH)
* Maternal known cardiac disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maternal hemodynamic parametrics changes (Cardiac Output, assessed by USCOM® system) in pregnancies complicated by congenital heart diseases and immediately after delivery | 36 months
  Hemodynamic indices will be obtained using the USCOM® system. Women will undergo a hemodynamic investigation at the time of first diagnosis of congenital heart disease during pregnancy or at the first assessment in Fondazione Policlinico A. Gemelli during pregnancy and then every two weeks until delivery. An additional hemodynamics evaluation will be performed in the post-partum period (in the 72 hours immediately after delivery). All hemodynamic assessment will be performed under standardized conditions. Heart rate (HR) and stroke volume will be combined to report cardiac output (CO) in L/min.
Maternal hemodynamic parametrics changes (Systemic vascular resistance, assessed by USCOM® system) in pregnancies complicated by congenital heart diseases and immediately after delivery | 36 months
  Hemodynamic indices will be obtained using the USCOM® system. Women will undergo a hemodynamic investigation at the time of first diagnosis of congenital heart disease during pregnancy or at the first assessment in Fondazione Policlinico A. Gemelli during pregnancy and then every two weeks until delivery. An additional hemodynamics evaluation will be performed in the post-partum period (in the 72 hours immediately after delivery). All hemodynamic assessment will be performed under standardized conditions. Systemic vascular resistance (dynes/s/cm5) will be evaluated.

SECONDARY OUTCOMES:
Prevalence of cases of preeclampsia in our population of pregnancies complicated by congenital heart disease | 36 months
  According to the International Society for the Study of Hypertension in Pregnancy (ISSHP) 2018 criteria, preeclampsia (PE) will be defined as de-novo hypertension (≥ 140/90 mmHg) after 20 weeks' gestation with coexisting proteinuria, other maternal organ dysfunction or fetal growth restriction.
Correlation between maternal hemodynamic profile (Cardiac Output) and perinatal outcome | 36 months
  Maternal hemodynamic indices will be obtained using the USCOM® system: heart rate (HR) and stroke volume will be combined to report cardiac output (CO) in L/min.
Correlation between maternal hemodynamic profile (Systemic vascular resistance) and perinatal outcome | 36 months
  Maternal hemodynamic indices will be obtained using the USCOM® system: systemic vascular resistance (dynes/s/cm5) will be evaluated.
Correlation between maternal hemodynamic profile and perinatal outcome (gestational age at delivery) | 36 months
  Perinatal outcome will be evaluated. Gestational age will be expressed as weeks and days at delivery.
Correlation between maternal hemodynamic profile and perinatal outcome (birthweight) | 36 months
  Perinatal outcome will be evaluated. Birthweight will be expressed in grams.
Correlation between maternal hemodynamic profile and perinatal outcome (birthweight centile) | 36 months
  Perinatal outcome will be evaluated. Birthweight centile will be expressed in centile.
Correlation between maternal hemodynamic profile and perinatal outcome (need of respiratory or cardiac support) | 36 months
  Perinatal outcome will be evaluated, such as need of respiratory or cardiac support.
Correlation between maternal hemodynamic profile and perinatal outcome (neonatal intensive care unit admission) | 36 months
  Perinatal outcome will be evaluated, such as neonatal intensive care unit admission.
Correlation between maternal hemodynamic profile and perinatal outcome (number of days in neonatal intensive care unit) | 36 months
  Perinatal outcome will be evaluated, such as number of days in neonatal intensive care unit.
Correlation between maternal hemodynamic profile and perinatal outcome (major neonatal complications) | 36 months
  Perinatal outcome will be evaluated, such as major neonatal complications.
Correlation coefficients between the maternal hemodynamic parameters (Cardiac output) to the specific heart defect type | 36 months
  The specific type of congenital heart defect, assessed using obstetric ultrasounds, will be related to maternal hemodynamic indices, assessed using the USCOM® system, such as Heart rate (HR) and stroke volume, combined to report cardiac output (CO) in L/min.
Correlation coefficients between the maternal hemodynamic parameters (Systemic vascular resistance) to the specific heart defect type | 36 months
  The specific type of congenital heart defect, assessed using obstetric ultrasounds, will be related to maternal hemodynamic indices, assessed using the USCOM® system, such as systemic vascular resistance (dynes/s/cm5).
Correlation coefficients between the maternal hemodynamic parameters (Cardiac output) to the specific fetal heart parameters | 36 months
  The specific fetal heart parameters (fetal cardiac function and morphologic features), assessed using obstetric ultrasounds, will be related to maternal hemodynamic indices, assessed using the USCOM® system, such as Heart rate (HR) and stroke volume, combined to report cardiac output (CO) in L/min.
Correlation coefficients between the maternal hemodynamic parameters (Systemic vascular resistance) to the specific fetal heart parameters | 36 months
  The specific fetal heart parameters (fetal cardiac function and morphologic features), assessed using obstetric ultrasounds, will be related to maternal hemodynamic indices, assessed using the USCOM® system, such as systemic vascular resistance (dynes/s/cm5).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Salvi, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome (Italy)
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Largo Francesco Vito 1, 00168, Rome (Italy), Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vinayagam D, Patey O, Thilaganathan B, Khalil A. Cardiac output assessment in pregnancy: comparison of two automated monitors with echocardiography. Ultrasound Obstet Gynecol. 2017 Jan;49(1):32-38. doi: 10.1002/uog.15915. PMID 26970353
- [Background] Hodgson LE, Venn R, Forni LG, Samuels TL, Wakeling HG. Measuring the cardiac output in acute emergency admissions: use of the non-invasive ultrasonic cardiac output monitor (USCOM) with determination of the learning curve and inter-rater reliability. J Intensive Care Soc. 2016 May;17(2):122-128. doi: 10.1177/1751143715619186. Epub 2015 Dec 10. PMID 28979476
- [Background] Brown MA, Magee LA, Kenny LC, Karumanchi SA, McCarthy FP, Saito S, Hall DR, Warren CE, Adoyi G, Ishaku S; International Society for the Study of Hypertension in Pregnancy (ISSHP). Hypertensive Disorders of Pregnancy: ISSHP Classification, Diagnosis, and Management Recommendations for International Practice. Hypertension. 2018 Jul;72(1):24-43. doi: 10.1161/HYPERTENSIONAHA.117.10803. No abstract available. PMID 29899139
- [Background] Melchiorre K, Giorgione V, Thilaganathan B. The placenta and preeclampsia: villain or victim? Am J Obstet Gynecol. 2022 Feb;226(2S):S954-S962. doi: 10.1016/j.ajog.2020.10.024. Epub 2021 Mar 24. PMID 33771361
- [Background] Masini G, Foo LF, Tay J, Wilkinson IB, Valensise H, Gyselaers W, Lees CC. Preeclampsia has two phenotypes which require different treatment strategies. Am J Obstet Gynecol. 2022 Feb;226(2S):S1006-S1018. doi: 10.1016/j.ajog.2020.10.052. Epub 2021 Jun 10. PMID 34774281
- [Background] Miremberg H, Gindes L, Schreiber L, Raucher Sternfeld A, Bar J, Kovo M. The association between severe fetal congenital heart defects and placental vascular malperfusion lesions. Prenat Diagn. 2019 Oct;39(11):962-967. doi: 10.1002/pd.5515. Epub 2019 Jul 17. PMID 31254468
- [Background] Thilaganathan B. Preeclampsia and Fetal Congenital Heart Defects: Spurious Association or Maternal Confounding? Circulation. 2017 Jul 4;136(1):49-51. doi: 10.1161/CIRCULATIONAHA.117.028816. No abstract available. PMID 28674092
- [Background] Boyd HA, Basit S, Behrens I, Leirgul E, Bundgaard H, Wohlfahrt J, Melbye M, Oyen N. Association Between Fetal Congenital Heart Defects and Maternal Risk of Hypertensive Disorders of Pregnancy in the Same Pregnancy and Across Pregnancies. Circulation. 2017 Jul 4;136(1):39-48. doi: 10.1161/CIRCULATIONAHA.116.024600. Epub 2017 Apr 19. PMID 28424221
- [Background] Auger N, Fraser WD, Healy-Profitos J, Arbour L. Association Between Preeclampsia and Congenital Heart Defects. JAMA. 2015 Oct 20;314(15):1588-98. doi: 10.1001/jama.2015.12505. PMID 26501535
- [Background] Brodwall K, Leirgul E, Greve G, Vollset SE, Holmstrom H, Tell GS, Oyen N. Possible Common Aetiology behind Maternal Preeclampsia and Congenital Heart Defects in the Child: a Cardiovascular Diseases in Norway Project Study. Paediatr Perinat Epidemiol. 2016 Jan;30(1):76-85. doi: 10.1111/ppe.12252. Epub 2015 Oct 19. PMID 26479038
- [Background] Llurba E, Sanchez O, Ferrer Q, Nicolaides KH, Ruiz A, Dominguez C, Sanchez-de-Toledo J, Garcia-Garcia B, Soro G, Arevalo S, Goya M, Suy A, Perez-Hoyos S, Alijotas-Reig J, Carreras E, Cabero L. Maternal and foetal angiogenic imbalance in congenital heart defects. Eur Heart J. 2014 Mar;35(11):701-7. doi: 10.1093/eurheartj/eht389. Epub 2013 Oct 24. PMID 24159191
- [Background] Taylor RN, Grimwood J, Taylor RS, McMaster MT, Fisher SJ, North RA. Longitudinal serum concentrations of placental growth factor: evidence for abnormal placental angiogenesis in pathologic pregnancies. Am J Obstet Gynecol. 2003 Jan;188(1):177-82. doi: 10.1067/mob.2003.111. PMID 12548214
- [Background] Hertig A, Berkane N, Lefevre G, Toumi K, Marti HP, Capeau J, Uzan S, Rondeau E. Maternal serum sFlt1 concentration is an early and reliable predictive marker of preeclampsia. Clin Chem. 2004 Sep;50(9):1702-3. doi: 10.1373/clinchem.2004.036715. No abstract available. PMID 15331514
- [Background] Levine RJ, Maynard SE, Qian C, Lim KH, England LJ, Yu KF, Schisterman EF, Thadhani R, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Circulating angiogenic factors and the risk of preeclampsia. N Engl J Med. 2004 Feb 12;350(7):672-83. doi: 10.1056/NEJMoa031884. Epub 2004 Feb 5. PMID 14764923
- [Background] Burton GJ, Woods AW, Jauniaux E, Kingdom JC. Rheological and physiological consequences of conversion of the maternal spiral arteries for uteroplacental blood flow during human pregnancy. Placenta. 2009 Jun;30(6):473-82. doi: 10.1016/j.placenta.2009.02.009. Epub 2009 Apr 17. PMID 19375795
- [Background] Abalos E, Cuesta C, Grosso AL, Chou D, Say L. Global and regional estimates of preeclampsia and eclampsia: a systematic review. Eur J Obstet Gynecol Reprod Biol. 2013 Sep;170(1):1-7. doi: 10.1016/j.ejogrb.2013.05.005. Epub 2013 Jun 7. PMID 23746796

DOCUMENTS (2):
  • Study Protocol (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT07092644/Prot_000.pdf
  • Informed Consent Form (2025-05-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT07092644/ICF_001.pdf